CLINICAL TRIAL: NCT02846532
Title: A Prospective, Open-Label, Active-Controlled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Efficacy of Rivaroxaban for Thromboprophylaxis in Pediatric Subjects 2 to 8 Years of Age After the Fontan Procedure
Brief Title: Pharmacokinetic, Pharmacodynamic, Safety, and Efficacy Study of Rivaroxaban for Thromboprophylaxis in Pediatric Participants 2 to 8 Years of Age After the Fontan Procedure
Acronym: UNIVERSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR108075; 39039039CHD3001 (Other: Janssen Research & Development, LLC); 2015-002610-76 (EudraCT Number)
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Results first posted 2022-03-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Thrombosis
Keywords: Thromboembolism; Fontan Procedure; Children
MeSH Terms: conditions — Thrombosis; Thromboembolism | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban
- Acetylsalicylic Acid (Experimental)
  Interventions: Drug: Acetylsalicylic Acid

INTERVENTIONS:
Drug: Rivaroxaban — Participants will receive oral suspension containing rivaroxaban 1 milligram per milliliter (mg/ml) twice daily in Part A and Part B. Following total daily doses of Rivaroxaban will be administered based on the weight of the participants: 7 to <8 kilogram (kg) will receive 2.2 milligram (mg); 8 to <10 kg will receive 3.2 mg; 10 to<12 kg will receive 3.4 mg; 12 to <20 will receive 4.0 mg and 20 to <30 will receive 5.0 mg.
  Arms: Rivaroxaban
Drug: Acetylsalicylic Acid — Participants will receive 5 milligram per kilogram (mg/kg) of acetylsalicylic acid once daily up to 12 months in Part B.
  Arms: Acetylsalicylic Acid

SUMMARY:
The Purpose of this study is to characterize the single and multiple-dose pharmacokinetic (PK) and pharmacokinetic/pharmacodynamic (PK/ PD) profiles after oral rivaroxaban therapy administered to pediatric participants 2 to 8 years of age with single ventricle physiology who have completed the Fontan procedure within 4 months prior to enrollment (Part A) and to evaluate the safety and efficacy of rivaroxaban, administered twice daily (exposure matched to rivaroxaban 10 milligram [mg] once daily in adults) compared to acetylsalicylic acid (ASA), given once daily (approximately 5 milligram per kilogram [mg/kg]) for thromboprophylaxis in pediatric participants 2 to 8 years of age with single ventricle physiology who have completed the Fontan procedure within 4 months prior to enrollment.

DETAILED DESCRIPTION:
Part A: This part includes a 12-day Initial PK, PD, and Safety Assessment Period. Participants in Part A will not participate in Part B. Randomization in Part B of this study will begin once the cumulative data from the Initial PK, PD, and Safety Assessment Period in Part A are deemed acceptable by the Independent Data Monitoring Committee. Part A of the study will consist of an up to 21-day Screening Period, a 12-day Initial PK, PD, and Safety Assessment Period, a 12-month Open-Label Treatment Period, and a 30-day Follow-Up phone contact. Part B: Participants will be randomly assigned to two treatment groups and randomization ratio will be 2:1 for rivaroxaban and ASA. ASA will be used as control. There will be an up to a 21-day Screening Period, a 12 month Open-Label Treatment Period and a 30-day Follow-Up phone contact.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be considered to be clinically stable by the investigator and able to tolerate oral or enteral administration of a suspension formulation and oral/enteral feedings
* Satisfactory initial post-Fontan transthoracic echocardiographic Screening as defined in the Post-Fontan Echocardiographic Examination Research Protocol
* Parent/legally acceptable representative must sign an informed consent form (ICF) and child assent will also be provided, if applicable, according to local requirements

Exclusion Criteria:

* Evidence of thrombosis, including those that are asymptomatic confirmed by post-Fontan procedure transthoracic echocardiogram, or other imaging techniques, during the Screening period of the study
* History of gastrointestinal disease or surgery associated with clinically relevant impaired absorption
* History of or signs/symptoms suggestive of protein-losing enteropathy
* Active bleeding or high risk for bleeding contraindicating antiplatelet or anticoagulant therapy, including a history of intracranial bleeding
* Platelet count less than (<)50*10^9/Liters (L) at Screening
* Estimated glomerular filtration rate (eGFR) <30 milliliters per minute per 1.73 meter square (mL/min/1.73m^2)
* Known clinically significant liver disease

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (42):
- United States (17):
  - Los Angeles, California
  - Gainesville, Florida
  - Oak Lawn, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Córdoba
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Brazil (3):
  - Curitiba
  - Porto Alegre
  - São Paulo
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Japan (4):
  - Fukuoka
  - Kitakyushu-shi
  - Setagaya Ku
  - Shizuoka
- Kuala Lumpur, Malaysia
- México, Mexico
- Netherlands (3):
  - Leiden
  - Rotterdam
  - Utrecht
- Spain (5):
  - A Coruña
  - Barcelona
  - Bilbao
  - Madrid
  - Valencia

REFERENCES:
- [Derived] McCrindle BW, Michelson AD, Van Bergen AH, Suzana Horowitz E, Pablo Sandoval J, Justino H, Harris KC, Jefferies JL, Miriam Pina L, Peluso C, Nessel K, Lu W, Li JS; UNIVERSE Study Investigators *. Thromboprophylaxis for Children Post-Fontan Procedure: Insights From the UNIVERSE Study. J Am Heart Assoc. 2021 Nov 16;10(22):e021765. doi: 10.1161/JAHA.120.021765. Epub 2021 Sep 24. PMID 34558312
- See also: ERF update upload receipt — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108075&attachmentIdentifier=ecc7606d-69c9-4747-8c64-2f0ad414eacd&fileName=2015-002610-76-_Receipt.png&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivaroxaban (Part A): Participants received rivaroxaban as 0.1 percent (%) (1 milligram per milliliter [mg/ml]) oral suspension with target exposure matching to that of rivaroxaban 10 mg given once daily in adults as per participant's body weight adjusted total daily dosing administered as two doses 12 hours apart (7 to less than [<] 8 kilograms [kg] participant received 2.2 mg; 8 to <10 kg received 3.2 mg; 10 to <12 kg received 3.4 mg; 12 to <20 kg received 4.0 mg; and 20 to <30 kg received 5.0 mg) (morning and evening dosing), up to 12 months.
- Rivaroxaban (Part B): Participants received rivaroxaban as 0.1% (1 mg/ml) oral suspension with target exposure matching to that of rivaroxaban 10 mg given once daily in adults as per participant's body weight adjusted total daily dosing administered as two doses 12 hours apart (7 to <8 kg participant received 2.2 mg; 8 to <10 kg received 3.2 mg; 10 to <12 kg received 3.4 mg; 12 to <20 kg received 4.0 mg and; 20 to <30 kg received 5.0 mg) (morning and evening dosing), up to 12 months.
- Aspirin (Part B): Participants received aspirin (acetylsalicylic acid) 5 mg/kg once daily up to 12 months.
Period: Overall Study
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B)
Started | 12 | 66 | 34
Completed | 11 | 63 | 33
Not Completed | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B) | Total
Number analyzed (Participants) | 12 | 66 | 34 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.5 (0.67) | 4.1 (1.74) | 4.2 (1.8) | 3.9 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 30 | 11 | 46
  Male | 7 | 36 | 23 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 22 | 11 | 34
  Not Hispanic or Latino | 11 | 42 | 19 | 72
  Unknown or Not Reported | 0 | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 14 | 7 | 21
  Black or African American | 3 | 8 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 8 | 40 | 20 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5
  Other | 1 | 2 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 5 | 1 | 6
  BELGIUM | 0 | 5 | 4 | 9
  BRAZIL | 0 | 7 | 10 | 17
  CANADA | 0 | 3 | 3 | 6
  JAPAN | 0 | 8 | 1 | 9
  MALAYSIA | 0 | 5 | 5 | 10
  MEXICO | 0 | 6 | 2 | 8
  NETHERLANDS | 0 | 1 | 0 | 1
  SPAIN | 5 | 1 | 0 | 6
  UNITED STATES | 7 | 25 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Thrombotic Event (Venous or Arterial and Symptomatic or Asymptomatic)
Description: Thrombotic event was defined as the appearance of a new thrombotic burden within the cardiovascular system on either routine surveillance or clinically indicated imaging, or the occurrence of a clinical event known to be strongly associated with thrombus (such as cardioembolic stroke, pulmonary embolism). The event included ischemic stroke, pulmonary embolism, venous thrombosis, arterial/intracardiac thrombosis, and other thrombosis.
Time Frame: Up to 12 months
Population: Full analysis set included all participants in Part A who received at least 1 dose of study drug and all participants in Part B who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B)
Number analyzed (Participants) | 12 | 64 | 34
percentage of participants
  Any thrombotic event | 8.3 | 1.6 | 8.8
  Ischemic stroke | 0 | 0 | 2.9
  Pulmonary embolism | 0 | 1.6 | 0
  Venous thrombosis | 8.3 | 0 | 5.9
  Arterial/intracardiac thrombosis | 0 | 0 | 0
  Other thrombosis | 0 | 0 | 0

2. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 1 (0.5-1.5 Hours Postdose)
Description: Plasma rivaroxaban concentrations for Parts A and B were assessed. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 0.5-1.5 hours postdose
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug and had quantifiable rivaroxaban plasma concentrations. Here, 'N' (number of participants analyzed) signifies number of participants that were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 60
micrograms per liter (mcg/L) | 46.69 (39.4) | 92.86 (72.6)

3. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 1 (1.5-4 Hours Postdose)
Description: as for outcome 2
Time Frame: Day 1: 1.5-4 hours postdose
Population: PK analysis set included all participants who received at least 1 dose of study drug and had quantifiable rivaroxaban plasma concentrations. Here, 'N' (number of participants analyzed) signifies number of participants that were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 61
mcg/L | 86.62 (43.1) | 103.61 (62.6)

4. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 4 (Up to 3 Hours Predose)
Description: as for outcome 2
Time Frame: Day 4: Up to 3 hours predose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
mcg/L | 36.58 (37.4) |

5. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 4 (0.5-1.5 Hours Postdose)
Description: as for outcome 2
Time Frame: Day 4: 0.5-1.5 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
mcg/L | 107.58 (54.2) |

6. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 4 (1.5-4 Hours Postdose)
Description: as for outcome 2
Time Frame: Day 4: 1.5-4 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
mcg/L | 147.18 (116) |

7. Primary Outcome: Plasma Concentration of Rivaroxaban at Day 4 (6-8 Hours Postdose)
Description: as for outcome 2
Time Frame: Day 4: 6-8 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
mcg/L | 66.81 (64.6) |

8. Primary Outcome: Plasma Concentration of Rivaroxaban at Month 3 (Up to 3 Hours Predose)
Description: as for outcome 2
Time Frame: Month 3: Up to 3 hours predose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 10 | 52
mcg/L | 38.23 (25.7) | 29.41 (25.5)

9. Primary Outcome: Plasma Concentration of Rivaroxaban at Month 3 (0.5-1.5 Hours Postdose)
Description: as for outcome 2
Time Frame: Month 3: 0.5-1.5 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 10 | 55
mcg/L | 86.25 (32.0) | 94.12 (82.2)

10. Primary Outcome: Plasma Concentration of Rivaroxaban at Month 3 (2.5-4 Hours Postdose)
Description: as for outcome 2
Time Frame: Month 3: 2.5-4 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 10 | 57
mcg/L | 96.67 (58.4) | 102.99 (56.0)

11. Primary Outcome: Percentage of Participants With Bleeding Events
Description: Bleeding events were categorized into major, clinically relevant non-major bleeding (CRNM), and trivial bleeding events. Major bleeding: overt bleeding and associated with a fall in hemoglobin of 2 gram per deciliter (g/dL) or more; or leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults; or occurring in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal; or contributing to death. CRNM bleeding: overt bleeding not meeting the criteria for major bleeding but associated with: Medical intervention, or Unscheduled contact with a physician, cessation of study treatment, or Discomfort for the subject such as pain, or Impairment of activities of daily life. Trivial bleeding: any other overt bleeding event that does not meet criteria for CRNM bleeding.
Time Frame: Up to 12 months
Population: Safety analysis set included all participants in Part A who received at least 1 dose of study drug and all participants in Part B who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B)
Number analyzed (Participants) | 12 | 64 | 34
percentage of participants
  Any bleeding event | 33.3 | 35.9 | 41.2
  Major Bleeding | 0 | 1.6 | 0
  Clinically relevant non-major bleeding | 8.3 | 6.3 | 8.8
  Trivial bleeding | 25.0 | 32.8 | 35.3

12. Primary Outcome: Absolute Prothrombin Time (PT) at Day 1 (0.5-1.5 Hours Postdose)
Description: Absolute prothrombin time was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 0.5-1.5 hours postdose
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug and had quantifiable and time-matched PT, activated partial thromboplastin time (aPTT), and/or anti-factor Xa (FXa) activity values were included in the descriptive PD analysis. Here, 'N' (number of participants analyzed) signifies number of participants that were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 56
seconds | 15.46 (1.90) | 18.02 (2.58)

13. Primary Outcome: Absolute PT at Day 1 (1.5-4 Hours Postdose)
Description: Absolute PT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 1.5-4 hours postdose
Population: PD analysis set included all participants who received at least 1 dose of study drug and had quantifiable and time-matched PT, aPTT, and/or anti-FXa activity values were included in the descriptive PD analysis. Here, 'N' (number of participants analyzed) signifies number of participants that were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 55
seconds | 16.58 (1.84) | 18.76 (2.25)

14. Primary Outcome: Absolute PT at Day 4 (Up to 3 Hours Predose)
Description: Absolute PT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average the participants included in the given time-range is presented here.
Time Frame: Day 4: Up to 3 hours predose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 15.21 (1.54) |

15. Primary Outcome: Absolute PT at Day 4 (0.5-1.5 Hours Postdose)
Description: as for outcome 13
Time Frame: Day 4: 0.5-1.5 hours postdose
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug and had quantifiable and time-matched PT, aPTT, and/or anti-FXa activity values were included in the descriptive PD analysis. Here, 'N' (number of participants analyzed) signifies number of participants that were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 17.95 (2.10) |

16. Primary Outcome: Absolute PT at Day 4 (1.5-4 Hours Postdose)
Description: as for outcome 13
Time Frame: Day 4: 1.5-4 hours postdose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 18.73 (3.30) |

17. Primary Outcome: Absolute PT at Day 4 (6-8 Hours Postdose)
Description: as for outcome 13
Time Frame: Day 4: 6-8 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 16.13 (2.13) |

18. Primary Outcome: Absolute PT at Month 3 (Up to 3 Hours Predose)
Description: as for outcome 13
Time Frame: Month 3: Up to 3 hours predose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 56
seconds | 17.59 (2.65) | 16.45 (2.27)

19. Primary Outcome: Absolute PT at Month 3 (0.5-1.5 Hours Postdose)
Description: as for outcome 13
Time Frame: Month 3: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 8 | 48
seconds | 20.13 (3.55) | 18.89 (3.69)

20. Primary Outcome: Absolute PT at Month 3 (2.5-4 Hours Postdose)
Description: as for outcome 13
Time Frame: Month 3: 2.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 7 | 51
seconds | 19.14 (2.61) | 19.69 (2.81)

21. Primary Outcome: Activated Partial Thromboplastin Time (aPTT) at Day 1 (0.5-1.5 Hours Postdose)
Description: aPTT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 56
seconds | 31.4 (4.68) | 30.69 (8.23)

22. Primary Outcome: aPTT at Day 1 (1.5-4 Hours Postdose)
Description: aPTT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 1.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 55
seconds | 32.83 (3.79) | 30.25 (3.80)

23. Primary Outcome: aPTT at Day 4 (Up to 3 Hours Predose)
Description: as for outcome 21
Time Frame: Day 4: Up to 3 hours predose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 33.08 (5.68) |

24. Primary Outcome: aPTT at Day 4 (0.5-1.5 Hours Postdose)
Description: aPTT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average the participants included in the given time-range is presented here.
Time Frame: Day 4: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 36.17 (6.99) |

25. Primary Outcome: aPTT at Day 4 (1.5-4 Hours Postdose)
Description: aPTT was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average for the participants included in the given time-range is presented here.
Time Frame: Day 4: 1.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 37.58 (8.45) |

26. Primary Outcome: aPTT at Day 4 (6-8 Hours Postdose)
Description: as for outcome 21
Time Frame: Day 4: 6-8 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 0
seconds | 32.83 (5.94) |

27. Primary Outcome: aPTT at Month 3 (Up to 3 Hours Predose)
Description: as for outcome 21
Time Frame: Month 3: Up to 3 hours predose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 12 | 51
seconds | 25.36 (3.76) | 28.70 (3.76)

28. Primary Outcome: aPTT at Month 3 (0.5-1.5 Hours Postdose)
Description: as for outcome 21
Time Frame: Month 3: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 8 | 48
seconds | 26.60 (2.55) | 31.15 (4.17)

29. Primary Outcome: aPTT at Month 3 (2.5-4 Hours Postdose)
Description: as for outcome 21
Time Frame: Month 3: 2.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 7 | 51
seconds | 26.74 (1.79) | 31.67 (3.58)

30. Primary Outcome: Anti-FXa at Day 1 (0.5-1.5 Hours Postdose)
Description: Anti-FXa was assessed as pharmacodynamic parameter. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here.
Time Frame: Day 1: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 6 | 43
mcg/L | 66.93 (23.9) | 99.46 (60.6)

31. Primary Outcome: Anti-FXa at Day 1 (1.5-4 Hours Postdose)
Description: as for outcome 30
Time Frame: Day 1: 1.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 11 | 52
mcg/L | 74.06 (32.4) | 104.57 (55.5)

32. Primary Outcome: Anti-FXa at Day 4 (6-8 Hours Postdose)
Description: as for outcome 30
Time Frame: Day 4: 6-8 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 11 | 0
mcg/L | 74.21 (60.6) |

33. Primary Outcome: Anti-FXa at Month 3 (Up to 3 Hours Predose)
Description: as for outcome 30
Time Frame: Month 3: Up to 3 hours predose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 3 | 17
mcg/L | 60.51 (29.4) | 53.41 (15.0)

34. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as those adverse events (AEs) that occurred from the first day of study drug to the last day of study drug + 2 days inclusive. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: Up to 12 months
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B)
Number analyzed (Participants) | 12 | 64 | 34
percentage of participants | 91.7 | 85.9 | 85.3

35. Primary Outcome: Anti-FXa at Month 3 (0.5-1.5 Hours Postdose)
Description: as for outcome 30
Time Frame: Month 3: 0.5-1.5 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 0 | 37
mcg/L |  | 110.90 (75.8)

36. Primary Outcome: Anti-FXa at Month 3 (2.5-4 Hours Postdose)
Description: as for outcome 30
Time Frame: Month 3: 2.5-4 hours postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B)
Number analyzed (Participants) | 0 | 51
mcg/L |  | 93.48 (50.3)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The safety population consisted of all participants in Part A who received at least 1 dose of study drug and all participants in Part B who were randomized and received at least 1 dose of study drug.
Arm/Group | Rivaroxaban (Part A) | Rivaroxaban (Part B) | Aspirin (Part B)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/64 | 0/34
Serious Adverse Events (participants affected / at risk) | 6/12 | 19/64 | 8/34
Other Adverse Events (participants affected / at risk) | 11/12 | 48/64 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Part A) (N=12) | Rivaroxaban (Part B) (N=64) | Aspirin (Part B) (N=34)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Periorbital Oedema (Eye disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Swelling Face (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Stoma Site Cellulitis (Infections and infestations) | 0 | 1 | 0
Vaccination Site Abscess (Infections and infestations) | 0 | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Wound Abscess (Infections and infestations) | 0 | 0 | 1
Stoma Site Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Investigation (Investigations) | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 0
Partial Seizures with Secondary Generalisation (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 2
Shock Haemorrhagic (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Part A) (N=12) | Rivaroxaban (Part B) (N=64) | Aspirin (Part B) (N=34)
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2
Gingival Bleeding (Gastrointestinal disorders) | 1 | 2 | 0
Tooth Loss (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 9 | 3
Pyrexia (General disorders) | 0 | 16 | 7
Bronchitis (Infections and infestations) | 2 | 3 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 5 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 3 | 1
Influenza (Infections and infestations) | 0 | 4 | 1
Nasopharyngitis (Infections and infestations) | 1 | 14 | 6
Otitis Media (Infections and infestations) | 0 | 4 | 3
Pharyngitis (Infections and infestations) | 0 | 5 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 5 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 9 | 5
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0
Viral Infection (Infections and infestations) | 2 | 2 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 5
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 4 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 6 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Haematoma (Vascular disorders) | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02846532/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT02846532/SAP_001.pdf